CLINICAL TRIAL: NCT05120102
Title: Influence of Low Level Laser Therapy on the Rate of Orthodontic Tooth Movement and Associated Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DuhsDikiohs
Record Dates: First submitted 2021-10-14; First posted 2021-11-15 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Orthodontic Appliance Complication
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental side of the arch (Experimental): The right or left side of the patients maxillary arch selected by randomization
  Interventions: Device: Diode laser
- Placebo side of the arch (No Intervention): The right or left side of the patients maxillary arch selected by randomization

INTERVENTIONS:
Device: Diode laser — K2 diode laser of 980nm wavelength
  Arms: Experimental side of the arch

SUMMARY:
This is a single blind randomized controlled trial with split mouth design including 45 patients with extractions of maxillary 1st bicuspids. First leveling and alignment will take place till 17 × 25 Stainless Steel wire pass passively through all the brackets. Canine retraction will be done through elastomeric ligatures maintaining force of 150gm on both sides. One of side of maxillary arch will be irradiated by diode laser (aluminum-gallium-arsenide) of 980nm on cervical, middle, and apical third on buccal and palatal surface of cuspid and the other side will act as placebo. Laser irradiation will be done at baseline and then for 3 more consecutive visits. Measurements will be recorded from maxillary canine hook to maxillary 1st molar hook at 3 weeks interval till complete canine retraction will be achieved. Patients will be given a questionnaires supported numeric scale to record their pain score for a week.

DETAILED DESCRIPTION:
First ethical approval for the study is going to be taken from the scientific committee and then Institutional Review Board of Dow University of Health Sciences. After getting informed consent from the chosen study participants, banding and bonding of the maxillary arch are going to be done through conventional fixed appliance Edgewise brackets. Initial leveling and alignment are going to be achieved by using nickel titanium and round stainless-steel wires until 0.017x0.025-inch stainless-steel wire passes passively through all fixed appliance. Anchorage is going to be implemented by skeletal anchorage through mini implants and molar stops on 0.017×0.025-inch stainless-steel wire just mesial to upper 1st molar band slot. As this study features a split mouth design so, every study subject will receive Gallium-Aluminum-Arsenic diode laser with a wavelength of 980nm ± 10nm on one maxillary canine and a placebo effect on the other maxillary canine. The side receiving laser irradiation is going to be alternated with every consecutive patient. To prevent from chauffeuring effect, a plastic shield will be used. The patient will be given questionnaire based scale to record pain score for a week.

Distalization of the canines is going to be accomplished by elastomeric chain (Medium span, Ortho Organizer) which can begin instantly after extraction of first premolars. There is no distinction between retraction rate of canines using either elastomeric chain or Nickel Titanium springs.

All study measurements will be taken using 0.01mm with digital Vernier caliper considering hook of maxillary cuspid teeth and hook of maxillary 1st molar teeth as reference points. Measurements will be recorded thrice in a single visit and mean is taken to avoid bias. Readings will be recorded after every three-weeks interval until one of the canines is completely retracted. Arch length will be measured on the cast as inter molar width. Patients will be given a questionnaire supported numeric scale to record their pain score for a week.

ELIGIBILITY:
Inclusion Criteria:

* age between 15-30 years
* Patients having symmetric extraction of maxillary 1st bicuspids
* All dentitions till 2nd molars should be erupted in the arch

Exclusion Criteria:

* Patients with Long term medication or with a history of radiotherapy or chemotherapy.
* Patients with Parafunctional habit.
* Patients with severe tooth displacement (ectopic canine), patients with missing teeth and impacted teeth (except third molars).
* Tooth morphological anomalies especially in the maxillary canines determined clinically or on OrthoPantomoGram/periapical X-rays.
* Patients with any systemic or metabolic disorder or bone pathology.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
orthodontic tooth movement | 6months
  tooth movement measured in millimeters

SECONDARY OUTCOMES:
orthodontic pain | 6months
  pain score through visual analogue scale having a score zero means no pain to score 5 means worst

CONTACTS AND LOCATIONS:
Overall Officials: Imtiaz Dr Ahmed, FCPS, Study Director — Supervisor
Locations (1):
- Dow university of health sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Visit duhs web page
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For a year after completion
Access Criteria: No such criteria
URL: http://duhs.edu.pk